CLINICAL TRIAL: NCT02098551
Title: Skin Testing With Recombinant Bet v 1 and Hypoallergenic Recombinant Bet v 1 Fragments to Dissect the Contribution of IgE to Chronic Allergic Skin Inflammation
Brief Title: Skin Testing With Recombinant Bet v 1 and Hypoallergenic Recombinant Bet v 1 Fragments
Status: Completed | Type: Observational
Sponsor: Stefan Woehrl (Other)
Collaborators: Medical University of Vienna (Other)
Responsible Party: Sponsor-Investigator, Stefan Woehrl, Mag. Dr. Stefan Wöhrl, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Other Study IDs: 147/2009
Record Dates: First submitted 2011-07-26; First posted 2014-03-28 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2015-12

CONDITIONS: Atopic Dermatitis
Keywords: atopic dermatitis; bet v 1; bet v 1 fragments; allergy
MeSH Terms: conditions — Dermatitis, Atopic; Hypersensitivity | interventions — APT

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Four (4): Group 1: Birch pollen-related atopic dermatitis (AD) (n=15) Group 2: Birch pollen allergic patients without AD (n=5) Group 3: Allergic individuals without birch pollen allergy (n=5) Group 4: Non-allergic individuals (n=5)
  Patients will be tested by SPT and APT:
  SPT: Histamine, buffer, commercial birch pollen extract, rBet v 1, rBet v 1 fragment 1, rBet v 1 fragment 2, and equimolar rBet v 1 fragment mix (20 and 40 μg/ml) in duplets.
  APT: birch pollen extract, rBet v 1, rBet v 1 fragment 1, rBet v 1 fragment 2, equimolar mix of rBet v 1 fragments (160 μg/application); negative control with vaseline
  Interventions: Other: SPT and APT

INTERVENTIONS:
Other: SPT and APT — All patients will be tested by skin prick testing (SPT: Histamine, buffer, commercial birch pollen extract, rBet v 1 (20 and 40 μg/ml), rBet v 1 fragment 1 (20 and 40 μg/ml), rBet v 1 fragment 2 (20 and 40 μg/ml), equimolar rBet v 1 fragment mix (20 and 40 μg/ml) in duplets.
  Atopy patch testing (APT: birch pollen extract, rBet v 1:160 μg/application, rBet v 1 fragment 1: 160 μg/application, rBet v 1 fragment 2: 160 μg/ml, equimolar mix of rBet v 1 fragments: 160 μg/application; negative control with vaseline alone.

SUMMARY:
Aim of this study is to use the major allergen 1 of birch-tree pollen (Bet v 1, Betula verrucosa, synonymous Betula pendula), to investigate the contribution of immunoglobulin E (IgE)- versus non-IgE-mediated mechanisms to chronic skin inflammation in atopic dermatitis patients.

DETAILED DESCRIPTION:
In this study non-IgE-reactive recombinant Bet v 1 (rBet v 1) fragments (F1: aa 1-74; F2: aa 75-160) and the fully IgE-reactive recombinant Bet v 1 (aa 1-160)will be used for skin prick testing and atopy patch testing in birch pollen allergic patients with birch pollen induced exacerbation of atopic dermatitis. For control purposes birch pollen allergic patients without birch pollen-induced atopic eczema, persons with allergies other than to birch and non-allergic people will be tested.

The individuals will be subjected to in vivo skin prick and atopy patch testing with rBet v 1, rBet v 1 fragment 1, rBet v 1 fragment 2 and an equimolar mix of the rBet v 1 fragments. In parallel, the IgE reactivity, and in vitro T cell proliferation, and cytokine production will be studied. Those analyses should help to determine the relevance of IgE mediated mechanisms to chronic skin inflammation and T cell proliferation in AD patients.

A staining for the surface markers chemokine receptor (CCR4)+ and cutaneous lymphocyte antigen (CLA)+ which reportedly are enriched in inflamed skin will further allow to investigate whether patients with high numbers of T lymphocytes expressing CCR4 and CLA tend to exhibit stronger skin inflammation. Moreover, allergen-specific antibody and T cell responses will be analyzed 6-8 weeks after the epicutaneous allergen application.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 75 years
2. They will be available to complete the study

Exclusion Criteria:

1. Severe general maladies
2. Severe skin inflammation in the test area
3. Risk of non-controllable general reaction
4. Pregnancy and breast-feeding
5. Autoimmune diseases, immune-defects including immuno-suppression, immune-complex-induced immunopathies
6. Contra-indication for adrenaline
7. Patients under long-term treatment with systemic corticosteroids immunosuppressive drugs, tranquilizers or psychoactive drugs
8. Positive IgE reaction on hypoallergenic Bet v 1 derivatives
9. The subject is currently participating in another clinical study in which the subject is or will be exposed to an investigational or a non-investigational drug.
10. The subject is at risk of non-compliance with the study procedures/restrictions

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Different types of individuals will be recruited and divided in four groups. A total of 30 allergic and non-allergic persons will be included in this study:
  patients with Birch pollen-related atopic dermatitis (AD), Birch pollen allergic patients without AD (group 2), allergic individuals without birch pollen allergy and non-allergic individuals.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2011-02; Primary Completion 2011-11 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Positive Atopy Patch Testing Reactions of Each Grade on the European Task Force on Atopic Dermatitis Scale | 6 months
  Birch pollen extract (BPE), as well as rBet v 1 (160mg), rBet v 1 fragment 1 (160mg), rBet v 1 fragment 2 (160mg), and an equimolar rBet v 1 fragment mix (80mg of each rBet v 1 fragment), were applied for 48h in patch test chambers onto nonlesional skin on the backs of the subjects. After 48h, patches were removed, and reactions were analyzed and photodocumented. Grading of positive APT reactions (i.e., reactions of more than 4 mm in diameter) was done according the European Task Force on Atopic Dermatitis by a blinded investigator: -, negative result; ?, only erythema, questionable; +, erythema, infiltration; ++, erythema, few papules (<3); +++, erythema, papules from 4 to less than many; ++++, erythema, many or spreading papules; or +++++, erythema, vesicles.

CONTACTS AND LOCATIONS:
Overall Officials: Rudolf Valenta, MD, Study Chair — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Result] Campana R, Moritz K, Marth K, Neubauer A, Huber H, Henning R, Blatt K, Hoermann G, Brodie TM, Kaider A, Valent P, Sallusto F, Wohrl S, Valenta R. Frequent occurrence of T cell-mediated late reactions revealed by atopy patch testing with hypoallergenic rBet v 1 fragments. J Allergy Clin Immunol. 2016 Feb;137(2):601-609.e8. doi: 10.1016/j.jaci.2015.08.042. Epub 2015 Oct 28. PMID 26518092